CLINICAL TRIAL: NCT01843114
Title: Measurement of Total Retinal Blood Flow in Patients With Diabetes and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-280113
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Type I Diabetes
Keywords: Retinal blood flow; Retinal vessel diameter; Fourier Domain Optical Coherence Tomography; Retinal blood velocities
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with Type I Diabetes (Other): 24 patients with type I diabetes with no or mild non-proliferative retinopathy
  Interventions: Device: FDOCT; Other: Dynamic Vessel Analyzer
- Healthy subjects (Other): 24 healthy age-and sex- matched control subjects
  Interventions: Device: FDOCT; Other: Dynamic Vessel Analyzer

INTERVENTIONS:
Device: FDOCT — Measurement of retinal blood velocities
  Other Names: Fourier Domain Color Doppler Optical Coherence Tomography
Other: Dynamic Vessel Analyzer — Measurement of retinal vessel diameters

SUMMARY:
The prevalence of diabetes and diabetes-associated complications is still increasing. Several major long-term complications of diabetes such as cardiovascular disease, chronic renal failure, diabetic retinopathy and others relate to the damage of blood vessels. Given that the eye provides the unique possibility in the human body to directly visualize blood vessels, much interest has been directed towards studying the ocular circulation. Although data of large epidemiological studies indicate that changes in retinal vessel caliber reflect other diabetes related factors, such as fasting glucose levels, there is still conflicting evidence on blood flow alterations in patients with diabetes. This is also related to the fact that up to now, methodological difficulties aggravate the assessment of blood flow changes in the retina in larger groups of patients. In the present study we propose to overcome this problem by using a technique called bi-directional Fourier Domain Doppler Optical Coherence Tomography (FDOCT), which we have developed in the recent years to measure retinal blood velocities. This technique allows for the non-invasive investigation of blood flow changes in human retina and will help us to better understand diabetes related vascular changes. The present study will use this technique to assess retinal blood flow changes in patients with diabetes and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects

* Men and women aged over 18 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt.

Inclusion criteria for patients with diabetes

* Men and women aged over 18 years
* Non-smokers
* Previously diagnosed type I diabetes
* No or mild non-proliferative diabetic retinopathy
* Normal ophthalmic findings except mild diabetic retinopathy, ametropia < 6 Dpt.

Exclusion Criteria:

Any of the following will exclude a healthy subject from the study:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptive)
* Arterial hypertension (defined as either systolic blood pressure >145 mmHg or diastolic blood pressure >90 mmHg)
* Blood donation during the previous three weeks
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropia >= 6 Dpt
* Pregnancy, planned pregnancy or lactating

Any of the following will exclude a patient with diabetes from the study:

* Participation in a clinical trial in the 3 weeks preceding the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition, except diabetes, as judged by the clinical investigator
* Arterial hypertension (defined as either systolic blood pressure >145 mmHg or diastolic blood pressure >90 mmHg)
* Blood donation during the previous three weeks
* Moderate to severe non-proliferative or proliferative diabetic retinopathy
* Previous laser photocoagulation treatment
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropia >= 6 Dpt
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Total retinal blood flow | 1 day
  Measurement of total retinal blood flow using the Dynamic Vessel Analyzer and Optical Coherence Tomography

SECONDARY OUTCOMES:
Retinal vessel diameter | 1 day
  Measurement of retinal vessel diameter using the Dynamic Vessel Analyzer
Retinal blood velocities | 1 day
  Measurement of retinal blood flow velocities using Fourier Domain Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Fondi K, Wozniak PA, Howorka K, Bata AM, Aschinger GC, Popa-Cherecheanu A, Witkowska KJ, Hommer A, Schmidl D, Werkmeister RM, Garhofer G, Schmetterer L. Retinal oxygen extraction in individuals with type 1 diabetes with no or mild diabetic retinopathy. Diabetologia. 2017 Aug;60(8):1534-1540. doi: 10.1007/s00125-017-4309-0. Epub 2017 May 25. PMID 28547132